CLINICAL TRIAL: NCT01967927
Title: Understanding GRID Radiation Therapy Effects on Human Tumor Oxygenation and Interstitial Pressure to Increase Translation of Solid Tumor Therapy
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study has been open for 8 years with no enrollment. Procedures in 2013 protocol are outdated. Cannot make the radiopharmaceutical on campus anymore.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 138725; 138725 (Other Grant/Funding Number: UAMS TRI)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: carcinoma; cancer; head; neck; otolaryngology
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma; Neoplasms | interventions — fluoromisonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GRID 18F-MISO (Experimental)
  Interventions: Drug: 18F-MISO

INTERVENTIONS:
Drug: 18F-MISO — A radiolabeled imaging agent that has been used for investigating tumor hypoxia with positron emission tomography (PET).
  Other Names: [18F]FMISO; [18F]FLUOROMISONIDAZOLE; 1H-1-(3-[18F]-FLUORO-2-HYDROXY-PROPYL)-2-NITRO-IMIDAZOLE

SUMMARY:
To estimate the mean and standard deviation (SD) of the post-treatment decreases in the interstitial fluid pressure and hypoxia-specific PET-scan signal from GRID-treated tumors in patients with locally advanced squamous-cell carcinoma of the head and neck.

The possible effects of GRID radiotherapy on tumor oxygenation levels and interstitial fluid pressure within the tumors will be measured by assessing the trend and statistical significance of the difference in values for each condition obtained prior to and just after GRID exposure in each subject enrolled in the study. We expect that there may be a trend for increases in tumor oxygenation and decreases in interstitial fluid pressure which would indicate that more accurately timed additional chemotherapy and radiation therapy would improve overall patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 80 years of age
* Karnofsky performance status greater than 70 or ECOG ≥ 2
* Cytological or histological documentation of squamous cell carcinoma of the head and neck, including the tongue, with a minimum tumor size of 6cm in any dimension.
* History of adequate hepatic function (endoscopic or percutaneous drainage as needed):

  a. AST (SGOT) / ALT (SGPT) ≤ 5X institutional ULN
* Chemotherapy naive
* History of adequate renal and bone marrow function:

  1. Leukocytes ≥ 3000/uL
  2. ANC ≥ 1500/uL
  3. Platelets ≥ 100000/UI
  4. Serum Creatinine ≤ 2.0 mg/dL

Exclusion Criteria:

* Women with a positive urine pregnancy test are excluded from this study; women of childbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to refrain from breast feeding and practice adequate contraception as specified in the informed consent. Adequate contraception consists of oral contraceptive, implantable contraceptives, injectable contraceptives, a double barrier method, or abstinence
* Subjects with active infections such as pneumonia, or wound infections that would preclude study procedures
* Subjects with known presence of central nervous system or brain metastases
* Subjects with prior radiotherapy to the head and neck region
* Subjects will be excluded if deemed unable to comply with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
To estimate the mean and standard deviation of the decrease in interstitial fluid pressure in tumors within 72 hours after GRID treatment. | within 72 hours after GRID treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Griffin, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States